CLINICAL TRIAL: NCT05195450
Title: TAF (Tenofovir Alafenamide) for Preventing Progression of Liver Disease in Non-cirrhotic Chronic HBV Infection With Normal ALT and Low Viral Load - a Randomized Controlled Trial
Brief Title: TAF (Tenofovir Alafenamide) for Preventing Progression of Liver Disease in Non-cirrhotic Chronic HBV Infection With Normal ALT and Low Viral Load.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HBV-02
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Non-cirrhotic, Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir Alafenamide Fumarate (Experimental): • TAF 25 mg OD vs no treatment x 5 years and beyond
  Interventions: Drug: Tenofovir alafenamide fumarate
- No Treatment Arm (No Intervention): No treatment

INTERVENTIONS:
Drug: Tenofovir alafenamide fumarate — • TAF 25 mg OD vs no treatment x 5 years and beyond
  Arms: Tenofovir Alafenamide Fumarate

SUMMARY:
The main goal of therapy for patients with chronic HBV infection with no significant liver disease is to improve survival and quality of life by preventing disease progression, development of liver cirrhosis and consequently HCC development. The likelihood of achieving these goals depends on the timing of therapy during the natural course of the infection but also on the stage of the disease and the patients' age when treatment is started. The inhibition of viral replication and normalization of ALT by antiviral treatment has been shown to achieve the elimination of chronic HBV-induced necroinflammatory activity and progressive fibrotic liver progression in the vast majority of patients, in turn reducing the risk of HCC. Even in HBeAg positive patients, treatment-induced HBeAg loss and seroconversion to antiHBe characterizes the induction of a partial immune control often leading to a low replicative phase of the chronic HBV infection and good outcomes.

Treatment in chronic HBV infection is indicated in - presence of advanced fibrosis/cirrhosis (LSM >11 KPA) or patients with significant fibrosis (LSM >8 or APRI >1.5 or >F2 on liver biopsy) with high viral load (>2000 IU/ml) or significantly elevated ALT (x2 ULN). Presence of any of these factors is known to increase the risk of development of cirrhosis and hepatocellular carcinoma. TAF in non-cirrhotic patients (LSM <8 KPA) with normal ALT and low viral load (HBV DNA <2000 IU/ml) (currently treatment ineligible) as compared to delayed initiation (on demand) might reduce HCC risk, progression of liver fibrosis and reduction in HBsAg levels. As TAF is known to have favorable effects on the overall long-term outcome, the main clinical challenge is to identify the patients at risk of HCC and cirrhosis who warrant early antiviral therapy.

DETAILED DESCRIPTION:
Aim and Objective - To study the safety and efficacy of TAF as compared to initiation based on current criteria in patients with non-cirrhotic chronic HBV infection and normal ALT and low viral load.

Methodology:

Study population: The study will be conducted on the treatment naïve consecutive patients having non-cirrhotic chronic HBV infection and normal ALT and low viral load seen at the outpatient clinics/wards of Department of Hepatology, ILBS, New Delhi.

Study design:

• A prospective, randomized, single center open label study.

Study period: 5 years from the last patient enrollment

Sample size with justification: All consecutive cases consenting to be a participant in this study and meeting inclusion and exclusion criteria will be enrolled. Considering the incidence of 20% for the composite end-point in patients without TAF and 5% for patients on TAF, with power of 80% and alpha error of 5%, 176 patients (88 patients in each arm) need to be enrolled. Considering the attrition rate of ~15%, we decide to enroll 100 patients in each arm.

Intervention

* TAF 25 mg OD vs no treatment x 5 years and beyond
* Tests - Baseline - USG abdomen, ALT, Creatinine, DEXA, HBVDNA, HBeAg, HBsAg (quant), Fibroscan
* 6 monthly - ALT
* 1 yearly - USG abdomen, ALT, Creatinine, DEXA, HBVDNA, HBeAg, HBsAg (quant), Fibroscan
* No liver biopsy

Statistical Analysis:

Data will be reported as mean + SD. Categorical variables will be compared using the chi-square test or Fisher exact test. Normal continuous variables will be compared using the Student's t test Non normal continuous variables will be compared using the Mann Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data). The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test. A Cox regression analysis will be performed to identify independent prognostic factors for survival. Univariate and multivariate analysis will be used whenever applicable.

Adverse effects:

Most common- headache, nausea, and fatigue; (1% to 10%): Abdominal pain, nausea, diarrhea, dyspepsia, elevated serum amylase, vomiting, flatulence, abdominal distension; Common (1% to 10%): Rash, pruritus, elevated ALT; Uncommon (0.1% to 1%): Treatment ALT flares.

ELIGIBILITY:
Inclusion Criteria:

- HBsAg+

* Persistent normal ALT 3-6m apart (<30 IU/ml in male and <20 IU/ml in female)
* HBV DNA < 2000 IU/ml
* LSM <8 Kpa

Exclusion Criteria:

* Prior NUC/IFN exposure
* Renal dysfunction (Serum Creatinine >1.5 mg/dl)
* Known liver cirrhosis/ esophageal varices
* Any clinical decompensation (CD)
* Pre-existing hepatocellular carcinoma
* Pregnancy
* Healthcare workers (HCW)
* Post transplant, patients with advance malignancy or on chemotherapy
* Co-infections - Hepatitis C, Hepatitis D, Human immunodeficiency virus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with HBV DNA <2000 IU/ml, normal ALT and no significant fibrosis (as per APASL 2015). | upto 5 Years
  Any two of the following -
  1. Significant fibrosis (LSM >8 Kpa or APRI >1.5)
  2. Persistently elevated ALT (2 consecutive ALT >30 U/ml 3-6m apart)
  3. HBV DNA >2000 IU/ml

SECONDARY OUTCOMES:
Incidence of HCC | upto 3 years
Incidence of HCC | upto 5 years
Percentage of patients with LSM >8 Kpa | upto 5 Years
Percentage of patients with LSM >11 Kpa | upto 5 Years
Number of subjects with no progression of fibrosis | upto 5 Years
Percentage of patients with APRI score >1.5 and >2 | upto 5 Years
Percentage of patients with HBV DNA >2000 IU/ml | upto 5 Years
Percentage of patients with undetectable HBV DNA | upto 5 Years
Percentage of patients with HBsAg loss and HBsAg seroconversion | upto 5 Years
Log HBsAg reduction | upto 5 Years
Percentage of patients with HBeAg loss and HBeAg seroconversion in HBeAg+ chronic hepatitis B | upto 5 Years
Percentage of patients with ALT > ULN, >2 times and 5 times ULN | upto 5 Years
Treatment related adverse effects of TAF | upto 5 Years
Non-compliant to treatment or monitoring | upto 5 years
Death | upto 5 years
Treatment related severe adverse effects | upto 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No